CLINICAL TRIAL: NCT03808441
Title: A Parallel Arm, Biomarker Driven, Phase II Trial to Determine the Role of Circulating Tumour DNA in Guiding a Switch Between Targeted Therapy and Immune Therapy in Patients With Advanced Cutaneous Melanoma
Brief Title: CAcTUS - Circulating Tumour DNA Guided Switch
Acronym: CAcTUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Bristol-Myers Squibb (Industry); University of Manchester (Other); Manchester Academic Health Science Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp129
Record Dates: First submitted 2018-11-07; First posted 2019-01-17 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Melanoma
Keywords: Circulating tumour DNA; targeted therapy; immune therapy; dabrafenib; trametinib; ipilimumab; nivolumab
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Arm (No Intervention): Dabrafenib + Trametinib
  Switch to N+I at first progression
- ctDNA Guided Switch (Active Comparator): Dabrafenib + Trametinib
  Switch to N+I when ctDNA levels in the blood have dropped by ≥80%.
  Interventions: Other: ctDNA analysis

INTERVENTIONS:
Other: ctDNA analysis — Regular ctDNA analysis, which upon a decrease in mutant BRAF VAF (variant allele frequency) level of ≥80% the switch to N+I is triggered.
  Arms: ctDNA Guided Switch

SUMMARY:
The stay aims to determine whether switching from targeted therapy to immunotherapy based on a decrease in levels of circulating tumour DNA in the blood, will improve the outcome in melanoma patients.

DETAILED DESCRIPTION:
The optimal scheduling of targeted and immune therapies in metastatic melanoma is unknown. At present, patients are treated with targeted therapy until acquired resistance develops, and then switched to immune therapy. Pre-clinical data has revealed that BRAF inhibition results in an environment that can enhance immune responses. Tumours responding to BRAF inhibitors but not resistant have been shown to have increased T cell infiltration, improved T cell recognition of melanoma associated antigens and reduced production of immunosuppressive cytokines. Furthermore, in response to targeted therapy LDH levels, which are associated with decreased response to immune therapy reduces, which may improve efficacy of immunotherapy.

A precise definition of response is required in order to decide upon a switch to immune therapy. A radiological definition of response is currently the standard assessment. However a scan at a fixed time point of 2 or 3 months does not reflect the wide range of response dynamics or allow decision making on an individual patient basis. The investigators have developed techniques using circulating tumour DNA (ctDNA) in the metastatic setting, which are able to accurately monitor tumour burden over time.

The aim of this pilot study is to provide a signal as to whether:

1. In BRAF mutant melanoma the efficacy of immune therapy is enhanced by response to pre-treatment with MAPK pathway inhibition with dabrafenib + trametinib.
2. Changes in ctDNA levels can be used to accurately inform when to switch from targeted to immune therapy.

Data from this study will provide the basis for follow on studies with sufficient power to assess whether tumours responding to BRAF inhibition as defined by response in ctDNA can improve efficacy of immune therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient capable of giving written informed consent
2. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
3. Histological confirmation of cutaneous melanoma
4. ≥ 16 years
5. Stage III un-resectable/ IV disease
6. BRAF p.V600E/K/R mutation confirmed (exact point mutation must be provided to the investigators)
7. At least one target lesion measurable by CT or MRI as per RECIST 1.1
8. Baseline ctDNA (as defined by the mutant BRAF VAF in plasma) ≥1.5%
9. Adequate organ function
10. ECOG performance status 0/1
11. Prior radiotherapy or radiosurgery must have been completed at least 2 weeks prior to the first dose of study drug
12. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
13. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drugs plus 5 half-lives of the drugs they are taking at treatment completion (5 times the half-life = 125 days [nivolumab]; 5 times the half-life = 90 days [ipilimumab]; 5 times the half life = 40 hours [dabrafenib]; 5 times the half life = 50 days [trametinib]) plus 30 days (duration of ovulatory cycle).
14. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment plus 5 half-lives of the study drug as above plus 90 days (duration of sperm turnover).
15. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements

Exclusion Criteria:

1. Prior systemic anti-cancer treatment (immune therapy, targeted therapy, vaccine therapy, or investigational treatment) for unresectable Stage III or Stage IV melanoma.
2. Prior adjuvant therapy with BRAF +/- MEK inhibitor or adjuvant therapy with combination PD-1 inhibitor plus CTLA-4 inhibitor. Prior adjuvant therapy with PD-1 inhibitor is allowed so long as relapse occurred > 6 months from discontinuation of treatment and treatment not stopped due to grade 3 or 4 toxicity.
3. Current use of a prohibited medication
4. History of another malignancy. Exception: patients who have been disease-free for 3 years, (i.e. patients with second malignancies that are indolent or definitively treated at least 3 years ago) or patients with a history of completely resected non-melanoma skin cancer. No additional therapy should be required whilst the patient is on study.
5. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the patients safety, obtaining informed consent, or compliance with study procedures.
6. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (patients with laboratory evidence of cleared or chronic (not active) HBV and HCV infection will be permitted).
7. A history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
8. Patients with active, known or suspected autoimmune disease. Patients with type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger will be permitted to enrol.
9. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
10. Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
11. Brain metastases and leptomeningeal metastases are excluded unless:

    * Asymptomatic and untreated at presentation, OR
    * Symptomatic lesions have been definitively treated with surgery or stereotactic surgery (whole-brain radiation may be given as adjuvant treatment), and do not require steroids for control of symptoms
    * Symptomatic metastases, treated or untreated, or metastases requiring steroids to control symptoms, are excluded
12. No enzyme inducing anticonvulsants for ≥ 4 weeks prior to randomisation
13. Coronary syndromes (including myocardial infarction within 6 months or unstable angina)
14. A history or evidence of current ≥ Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines with an ejection fraction of <50%
15. Treatment refractory hypertension defined as a blood pressure of systolic> 150 mmHg and/or diastolic > 95 mm Hg on >3 occasions which cannot be controlled by anti-hypertensive therapy;
16. Known cardiac metastases;
17. Uncorrectable electrolyte abnormalities (e.g. hypokalaemia, hypomagnesaemia, hypocalcaemia), long QT syndrome or taking medicinal products known to prolong the QT interval.
18. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes)
19. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments including monoclonal antibodies, their excipients, and/or dimethyl sulfoxide (DMSO) and/or Polysorbate-80-containing infusions.
20. Females who are breast-feeding.
21. Prisoners or patients who are involuntarily incarcerated.
22. Patients who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
CtDNA result critical (red) blood samples returned within 7 working days of samples being received in the laboratory | 12 months from last patient starting trial treatment
  Feasibility of returning samples to hospitals from the laboratory to inform clinical decisions
Decrease in ctDNA level of mutant BRAF≥80% | Through study completion, an average of 1 year
  To assess whether a decrease in ctDNA levels of mutant BRAF by ≥80% on targeted therapy is an appropriate cut off for switching to immune therapy

SECONDARY OUTCOMES:
Screen failure due to ctDNA levels of mutant BRAF VAF <1.5% Efficacy | Through study completion, an average of 1 year
  To assess whether BRAF VAF (within the ctDNA) of ≥1.5% is an appropriate target for study inclusion (by assessing the number and proportion of screen failures
First progression free survival (PFS) at 12 months | Through study completion, an average of 1 year
  To explore whether PFS at 12 months would improve in patients switching from targeted to immune therapy on response to treatment as guided by ctDNA levels of mutant BRAF VAF
First progression free survival | When all patients finished follow up, 4 years after last patient starting treatment
  Time to first progression in both arms
Second progression free survival | When all patients finished follow up, 4 years after last patient starting treatment
  Time to second progression in both arms
Overall survival | When all patients finished follow up, 4 years after last patient starting treatment
  Explore whether survival outcomes would improve in patients switching from targeted to immune therapy on response to treatment as guided by ctDNA levels of mutant BRAF VAF

OTHER OUTCOMES:
Time to ctDNA first progression | Through study completion, an average of 1 year
  Time to first progression measured by ctDNA
Time to ctDNA second progression | Through study completion, an average of 1 year
  Time to second progression measured by ctDNA
Increase in ctDNA levels of BRAF VAF during washout period from targeted to immune therapy switch in arm B | When all patients finished treatment, an average of 1 year after last patient starting treatment
Duration of mutant BRAF VAF (within ctDNA) response to targeted therapy | When all patients finished treatment, an average of 1 year after last patient starting treatment
Duration of mutant BRAF VAF (within ctDNA) response to immune therapy | When all patients finished treatment, an average of 1 year after last patient starting treatment
Time between observing rise in ctDNA levels of mutant BRAF VAF and progressive disease observed on scheduled scan | When all patients finished treatment, an average of 1 year after last patient starting treatment
  To explore the relationship between observing a rise in ctDNA level of mutant BRAF VAF and progressive disease observed from scheduled scan results
Time taken for mutant ctDNA level of mutant BRAF VAF to reach ≥80% decrease on targeted therapy | When all patients finished treatment, an average of 1 year after last patient starting treatment
  To compare duration in ctDNA level of mutant BRAF VAF response to targeted therapy between study arms
ctDNA level of mutant BRAF VAF (at each follow-up assessment timepoint) | When all patients finished treatment, an average of 1 year after last patient starting treatment
  To compare duration in ctDNA level of mutant BRAF VAF (within ctDNA) response to immune therapy between study arms
Best overall response rate to immune therapy | hen all patients finished treatment, an average of 1 year after last patient starting treatment
  To explore whether switching from targeted to immune therapy on treatment response as guided by ctDNA levels of mutant BRAF VAF will increase response to therapy
Duration of response to immune therapy | When all patients finished treatment, an average of 1 year after last patient starting treatment
Progression free survival on immune therapy from date of commencement of immune therapy | When all patients finished treatment, an average of 1 year after last patient starting treatment
  Time to progression on immune therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lorigan, Principal Investigator — The Christie National Health Service (NHS) Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No